CLINICAL TRIAL: NCT00492934
Title: Natural Cycle Versus Stimulation With Human Menopausal Gonadotropin in Cycles With Cryopreserved Embryos
Brief Title: What is the Best Preparation for Embryo Transfer in Cryo Cycles: a Natural Cycle or Light Hormonal Stimulation?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Thomas D'Hooghe, Professor, Medical Doctor, University Hospital, Gasthuisberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML2436 - 30/12/2003
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Infertility
Keywords: subfertility; endometrium thickness; implantation rate; embryo cryopreservation; embryo transfer
MeSH Terms: conditions — Infertility | interventions — Menotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Daily injections with a small dose of gonadotrophins from day 2 of the cycle
  Interventions: Drug: human menopausal gonadotrophins
- 2 (No Intervention): No daily injections with hormones

INTERVENTIONS:
Drug: human menopausal gonadotrophins — Daily subcutaneous injections, dose 37.5 IU or 75 IU, start on day 2 of the menstrual cycle until ovulation
  Other Names: Menopur
  Arms: 1

SUMMARY:
The study investigates if, among women with a regular cycle (between 25 and 45 days), the endometrium is better prepared for the transfer of an embryo that was cryopreserved and if the subsequent embryo implantation rate is higher when the cycle is started with daily, small-dose hormonal injections than in cycles without these daily injections.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Women with a regular cycle (between 21 and 35 days).
* Embryos with 50% intact blastomeres after thawing.
* Embryo and endometrium are synchronized.

Exclusion Criteria:

* Embryo storage time not longer than 5 years.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2004-01; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
implantation rate per embryo | 15 days after the embryo transfer

SECONDARY OUTCOMES:
thickness of the endometrium | 0-2 days before the human chorionic gonadotropin (hCG) injection

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D'Hooghe, MD, PhD, Study Director — University Hospital Gasthuisberg, Catholic University Leuven, Belgium
Locations (1):
- Leuven University Fertility Center, Leuven, Vlaams Brabant, Belgium

REFERENCES:
- [Derived] Peeraer K, Couck I, Debrock S, De Neubourg D, De Loecker P, Tomassetti C, Laenen A, Welkenhuysen M, Meeuwis L, Pelckmans S, Meuleman C, D'Hooghe T. Frozen-thawed embryo transfer in a natural or mildly hormonally stimulated cycle in women with regular ovulatory cycles: a RCT. Hum Reprod. 2015 Nov;30(11):2552-62. doi: 10.1093/humrep/dev224. Epub 2015 Sep 12. PMID 26364081